CLINICAL TRIAL: NCT04987827
Title: Investigating the Clinical Features and Prognosis of Bronchiectasis Adult Patients: a Multi-center, Primary Data, Cohort Study (ICON)
Brief Title: Investigating the Clinical Features and Prognosis of Bronchiectasis Adult Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ICON
Record Dates: First submitted 2021-07-09; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Bronchiectasis Adult
Keywords: Bronchiectasis; Non-Interventional Study
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bronchiectasis is a chronic respiratory disease characterized by permanent bronchiectasis.The incidence and prevalence of bronchiectasis have assumed continuously grows in global. Different from overseas, bronchiectasis is common disease in China. This study will collect data from the real-world bronchiectasis database and follow up for one year, describe the bronchiectasis exacerbation rate and proportions for frequent exacerbation, clinical features and prognosis of bronchiectasis exacerbation, the treatment pattern (when clinically stable) during follow-up period; and describe characteristics of bronchiectasis at baseline. This study will also explore potential baseline risk factors for bronchiectasis exacerbation during follow-up period.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic respiratory disease characterized by permanent bronchiectasis, its main clinical symptoms are cough, dyspnea, hemoptysis and recurrent respiratory tract infections. The incidence and prevalence of bronchiectasis have assumed continuously grows in global. Different from overseas, bronchiectasis is common disease in China. In 2013, the prevalence rate of bronchiectasis in Chinese residents over 40 years old was 1,200/100,000. As lack of large epidemiological data in China, the prevalence rate may still be underestimated, which needs more attention and research.

Bronchiectasis has heavy disease burden, characterized by recurrent acute exacerbations, high mortality, poor prognosis and heavy economic burden. The key points of bronchiectasis treatment strategy include exacerbation prevention, number of exacerbations reduction, prognosis improvement and then the quality of patients' life improvement. Therefore, it is important to describe the clinical features and prognosis of bronchiectasis (especially the incidence of acute exacerbations and the proportion of frequent exacerbations), and it would be helpful to understand the characteristics of bronchiectasis and standardize related diagnosis and treatment strategy.

This study will collect data from the real-world bronchiectasis database and follow up for one year, describe the bronchiectasis exacerbation rate and proportions for frequent exacerbation, clinical features and prognosis of bronchiectasis exacerbation, the treatment pattern (when clinically stable) during follow-up period; and describe characteristics of bronchiectasis at baseline. This study will also explore potential baseline risk factors for bronchiectasis exacerbation during follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bronchiectasis (according to the Chinese consensus, patient's previous chest CT examination must show bronchiectasis).
* Patients with age ≥18 years old.

Exclusion Criteria:

* Bronchiectasis due to known cystic fibrosis.
* With acute bronchiectasis exacerbation within 4 weeks before enrolment.
* Participated in any interventional clinical trial within 6 months before enrolment.
* Patients who are unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is designed that from 2021 Q4 to 2022 Q2, 1,250 bronchiectasis patients will be enrolled from 30 participating sites in China.
  *Bronchiectasis exacerbation defined as patients have three or more of the following six symptoms including cough, expectoration, purulent sputum, dyspnoea, fatigue, haemoptysis, and these symptoms persist more than 48 hours, and physicians prescribe systemic antibiotics due to these symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Bronchiectasis exacerbation times | one year
  Bronchiectasis exacerbation times (per person per year) during one year follow up.

SECONDARY OUTCOMES:
Proportions of different bronchiectasis exacerbations | one year
  Proportions of different bronchiectasis exacerbations(0, 1, 2, 3, ≥4 exacerbations per person per year) during one year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No